CLINICAL TRIAL: NCT05427370
Title: The Canadian CABG or PCI in Patients With Ischemic Cardiomyopathy Trial
Brief Title: The Canadian CABG or PCI in Patients With Ischemic Cardiomyopathy Trial (STICH3C)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sunnybrook Health Sciences Centre (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); Weill Medical College of Cornell University (Other)
Responsible Party: Principal Investigator, Stephen E. Fremes, Professor of Surgery, University of Toronto, Sunnybrook Health Sciences Centre
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: v.1.6; August 22, 2025
Record Dates: First submitted 2022-06-08; First posted 2022-06-22 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Coronary Artery Disease; Heart Failure Systolic
Keywords: Left ventricular dysfunction; CABG; PCI; MACCE
MeSH Terms: conditions — Coronary Artery Disease; Heart Failure, Systolic; Ventricular Dysfunction, Left

STUDY DESIGN:
Intervention Model Description: The STICH3C trial is a prospective, unblinded, international multi-center randomized trial of comparing revascularization by PCI vs. CABG in patients with multivessel/LM CAD and reduced LVEF.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Revascularization by PCI (Experimental): Revascularization will be attempted on/for significant lesions in major coronary vessels/side branches as planned by the local Heart Team, with the general recommendation of stenotic/occluded vessels with diameter >2.0 mm for PCI. The Heart Team consists of a minimum of one heart failure cardiologist, one interventional cardiologist and one cardiac surgeon.
  Interventions: Procedure: Revascularization by PCI
- Revascularization by CABG (Experimental): Revascularization will be attempted on/for significant lesions in major coronary vessels/side branches as planned by the local Heart Team, with the general recommendation of stenotic/occluded vessels with diameter >1.5 mm for CABG. The Heart Team consists of a minimum of one heart failure cardiologist, one interventional cardiologist and one cardiac surgeon
  Interventions: Procedure: Revascularization by CABG

INTERVENTIONS:
Procedure: Revascularization by PCI — Contemporary, "State-of-the-art" PCI techniques will be encouraged in STICH3C, based on the most recent evidence and clinical practice guidelines recommendations. The best practices to be followed include the use of physiological and intravascular guidance, new-generation drug-eluting stents or scaffolds, rotational or orbital atherectomy for extensive calcifications, recommended bifurcation techniques, chronic total occlusion for viable segments by experienced operators, and trans-radial access.Planned temporary ventricular support is permitted by experienced operators when deemed indicated.
  Arms: Revascularization by PCI
Procedure: Revascularization by CABG — The surgical revascularization strategy will be tailored according to the individual patient's coronary anatomy, left ventricular remodeling, aortic atherosclerosis, co-morbidities, local expertise, and surgical judgement. An internal thoracic artery will be used to graft the left anterior descending in all cases. Multi-arterial grafting may be considered in patients without significant co-morbidities and with expected limited vasopressor use, or in patients without saphenous conduits. Choice of on- vs. off-pump surgery is influenced by LV size, associated valvular disease, and aortic atherosclerosis, as well as surgeon experience, but on-pump surgery is recommended routinely. The use of adjunctive intra-aortic balloon support or other cardiac support is not routinely recommended in stable patients; the intra-aortic balloon support is the first line mechanical support.
  Arms: Revascularization by CABG

SUMMARY:
The Canadian CABG or PCI in Patients With Ischemic Cardiomyopathy (STICH3C) trial is a prospective, unblinded, international multi-center randomized trial of 754 subjects enrolled in approximately 45 centers comparing revascularization by percutaneous coronary intervention (PCI) vs. coronary artery bypass grafting (CABG) in patients with multivessel/left main (LM) coronary artery disease (CAD) and reduced left ventricular ejection fraction (LVEF).

The primary objective is to determine whether CABG compared to PCI is associated with a reduction in all-cause death, stroke, spontaneous myocardial infarction (MI), urgent repeat revascularization (RR), or heart failure (HF) readmission over a median follow-up of 5 years in patients with multivessel/LM CAD and ischemic left ventricular dysfunction (iLVSD).

Eligible patients are considered by the local Heart Team appropriate and amenable for non-emergent revascularization by both modes of revascularization.

The secondary objectives are to describe the early risks of both procedures, and a comprehensive set of patient-reported outcomes longitudinally.

DETAILED DESCRIPTION:
The evidence comparing PCI and CABG with medical therapy in patients with iLVSD has been the subject of multiple systematic reviews/meta-analyses of observational studies with inconsistent results. There is a current lack of evidence from properly powered randomized trials comparing contemporary state-of-the-art PCI vs. CABG to guide the clinical management in the vulnerable population of patients with iLVSD. Understanding the relative impact of both revascularization strategies on clinical outcomes in this prevalent population would have important clinical implications.

The overarching aim of the STICH3C trial is to compare the clinical efficacy and safety of contemporary PCI and CABG to treat patients with multivessel/left main (LM) CAD and iLVSD.

Participants will be allocated in a 1:1 ratio to either study arm using permuted block randomization stratified for study center and acute coronary syndrome (ACS) presentation through a centrally controlled, automated, web system. Eligible patients who provide informed consent can be enrolled. It is expected that initial revascularization will take place within 2 weeks of randomization. Staged PCI is expected to take place within 90 days of randomization. The recruitment will occur over 3 years, with a total study duration of 7 years, and a median duration of follow-up of 5 years.

ELIGIBILITY:
Inclusion Criteria:

1. Age >18 years;
2. LVEF ≤40% quantified by either echocardiography, SPECT ventriculography, or magnetic resonance within 2 months of randomization;
3. Prognostically important multivessel CAD (triple vessel CAD or double vessel disease including the left anterior descending (LAD) or LM). Significant coronary stenosis is defined as ≥ 70% based on coronary angiography, and/or fractional flow reserve (FFR) ≤0.80 or instantaneous wave-free ratio (iFR) ≤0.89. For LM disease, significant coronary stenosis is defined as >50% based on coronary angiography, intravascular ultrasound (IVUS) minimal luminal area (MLA) ≤6.0 mm2 (<4.5 mm2 Asian descent), or equivalent optical coherence tomography (OCT) measurements;
4. The institutional Heart Team agrees that guideline-directed medical therapy (GDMT) has been initiated for ≥1 month in prevalent and newly diagnosed cases. In patients hospitalized with newly diagnosed iLVSD (with or without acute coronary syndrome (ACS)) requiring revascularization before discharge, GDMT needs to be initiated, when possible in-hospital before randomization, with the expectation that it will be titrated to maximally tolerated doses after revascularization;
5. Signed informed consent.

Exclusion Criteria:

1. Decompensated HF requiring inotropic/adrenergic support, invasive or non-invasive ventilation or intra-aortic balloon pump/ventricular assist device therapy less than 48 hours prior to randomization;
2. Recent (<4 weeks) ST-elevation MI;
3. Concomitant severe valvular disease or other condition such as left ventricular aneurysm requiring surgical repair or replacement;
4. Planned major concomitant surgical procedures (LAAO and AF ablation surgical procedures permitted);
5. Prior PCI within the past 12 months (to reduce restenosis events from prior PCIs contributing to the primary outcome);
6. Prior cardiac surgery;
7. Prohibitive bleeding risk mandating avoidance of dual antiplatelet therapy;
8. Circumstances likely to lead to poor treatment adherence;
9. Severe end-organ dysfunction (such as dialysis, liver failure, respiratory failure, cancer) that reduces life expectancy to less than 5 years;
10. Current pregnancy;
11. Patient not amenable to both CABG or PCI according to the Heart Team;
12. Takotsubo/Takotsubo Cardiomyopathy/Broken Heart Syndrome.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 754 (Estimated)
Dates: Start 2023-06-22 (Actual); Primary Completion 2029-04 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
The Primary outcome is a Composite of all-cause mortality, stroke, spontaneous myocardial infarction, urgent repeat revascularization or heart failure readmission. | Median follow-up of 5 years.
  Time to event outcome measured as the time from randomization to the occurence of the first event.

SECONDARY OUTCOMES:
Death | At 30 days , 90 days and through study completion with a median follow-up of 5 years.
  Death will be reported at 30 days. Death over the entire duration of study will be reported as a time to event outcome. Death will be adjudicated as cardiovascular, non-cardiovascular and unknown.
Myocardial Infarction (MI) | At 30 days and through study completion with a median follow-up of 5 years.
  Periprocedural/perioperative MI is defined as <48 hours from revascularization. Spontaneous MI is defined as > or = 48 hours post revascularization
Number of participants with Stroke | At 30 days , 90 days and through study completion with a median follow-up of 5 years.
  Strokes will be classified as ischemic, hemorrhagic or uncertain.
Repeat Revascularization (RR) | At 30 days , 90 days and through study completion with a median follow-up of 5 years.
  Only urgent clinically driven unplanned repeat revascularizations by either PCI or CABG count towards primary ouctome. RR will be classified according to type (CABG vs. PCI), by location (target vessel vs. target lesion vs. graft vs. other), and whether clinically vs. non-clinically driven. Stent thrombosis (ARC defined) and graft thrombosis/ occlusion will be reported.
Hospitalizations | Through study completion with a median follow-up of 5 years.
  Hospitalizations will be defined as cardiac or non-cardiac. Hospitalizations will be reported as the number of participants with hospitalizations and as a count.
Composite of death/stroke/spontaneous MI | Through study completion with a median follow-up of 5 years.
  Measured as a time-to-event.
Composite of death/stroke/spontaneous MI/RR | Through study completion with a median follow-up of 5 years.
  Measured as a time-to-event.
Composite of death or cardiac hospitalization | Through study completion with a median follow-up of 5 years.
  Measured as a time-to-event.
Coronary composite endpoint | Through study completion with a median follow-up of 5 years.
  Coronary heart disease death, non-fatal MI, and coronary revascularization procedure. Measured as time-to-event outcome.
Heart Failure endpoint | Through study completion with a median follow-up of 5 years.
  Heart Failure Event (composite of heart failure death, heart failure hospitalization or revascularization for HF). Measured as time-to-event outcome.
Hierarchal Heart Failure outcome | Through study completion with a median follow-up of 5 years.
  The key hierarchal outcome of time to death and frequency of HF rehospitalizations will be tested using a win ratio
Number of participants with advanced Heart failure therapies | Through study completion with a median follow-up of 5 years.
  This includes - ICD/CRT implantation,Mitral valve repair (transcatheter/surgical),Ventricular Assist Device and Heart Transplant
Major Adverse Events | Results will be reported at 30 days and 90 days after index procedure (and 30 days after any planned staged PCI, allowed up to 90 days after randomization) as cardiac surgical hospitalizations maybe prolonged.
  These will be reported as the composite and individually: new renal replacement therapy, major bleeding (Bleeding Academic Research Consortium (BARC) 3-5), major vascular complication (according to VARC-2 criteria), unplanned RR, other reoperation, surgical site complication, intubation >48 hours, cardiac arrest, advanced cardiac life support, stroke and death.

OTHER OUTCOMES:
Kansas City Cardiomyopathy Questionnaire-12 | Through study completion with a median follow-up of 5 years.
  The scores range from 0-100 with higher scores indicating higher quality of life. The scores are classified as 0 to 24: very poor to poor; 25 to 49: poor to fair; 50 to 74: fair to good; and 75 to 100: good to excellent.
Seattle Angina Questionnaire-7 | Through study completion with a median follow-up of 5 years.
  It generates a summary score (scale 0-100, 100 = full health, 0 = worst health).
Short Form 12 Questionnaire | Through study completion with a median follow-up of 5 years.
  Scores range from 0 to 100, with higher scores indicating better physical and mental health functioning.
EuroQol-5D (EQ-5D) | Through study completion with a median follow-up of 5 years.
  Each dimension in the EQ-5D-5L has five response levels: no problems (Level 1); slight; moderate; severe; and extreme problems (Level 5). The EQ-5D index score is anchored at 1 (full health) and 0 (death).
Montreal Cognitive Assessment (MoCA) | Through study completion with a median follow-up of 5 years.
  Scores on the MoCA range from 0-30; a score of 26 or above is considered normal with higher scores indicating higher cognitive function.
Composite of severe stroke/ventilator dependance/new onset or worsening heart failure/ nursing home admission/ or new onset dialysis | Reported at 1 and 5 years and as a cumulative incidence.
  It will be measured as a time to event outcome.
Composite of stroke, nursing home admission and 3 or more non-elective admissions per 12 months | Reported at 1 and 5 years and as a cumulative incidence.
  It will be measured as a time to event outcome.
Length of stay outcomes | Reported at 90 days, 1 year and 5 years - this is only for DAOH.
  Length of stay of index ICU admission, Length of hospital stay of index admission. Days alive and out of hospital (DAOH).
Cumulative costs | 4 years.
  Cumulative costs will be collected over 4 years.
Cost-effectiveness | 4 years.
  Quality adjusted life years over four years based on EQ-5D at each follow-up time point and four-year cumulative costs.

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Fremes, MD,MSc,FRCSC, Principal Investigator — Sunnybrook Health Sciences Center, Toronto, Canada; Mario Gaudino, MD,PhD, Principal Investigator — Weill Medical College of Cornell University, USA; Jean L Rouleau, MD,PhD, Principal Investigator — Montreal Heart Institute, QC Canada; Guillaume Maquis-Gravel, MD,MSc, Principal Investigator — Montreal Heart Institute, QC Canada
Locations (40):
- United States (6):
  - Cedars-Sinai, Los Angeles, California
  - Yale University, New Haven, Connecticut
  - UofL Health, Inc, Louisville, Kentucky
  - John Hopkins Hospital, Baltimore, Maryland
  - Mayo Clinic, Rochester, Minnesota
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
- Medical University of Vienna, Vienna, Austria
- Heart Institute, Medical School of the University of Sao Paulo_INCOR, São Paulo, Brazil
- Canada (16):
  - University of Calgary; Libin Cardiovascular Institute, Calgary, Alberta
  - Mackenzie Health Sciences Center, Edmonton, Alberta
  - Fraser Health; Royal Columbian Hospital, New Westminster, British Columbia
  - Providence Health, Vancouver, British Columbia
  - Queen Elizabeth II Hospital, Halifax, Nova Scotia
  - Hamilton General Hospital, Hamilton, Ontario
  - London Health Sciences Center, University Hospital, London, Ontario
  - Southlake Regional HC, Newmarket, Ontario
  - Ottawa Heart Institute, Ottawa, Ontario
  - Sunnybrook Health Sciences Center, Toronto, Ontario
  - St. Michael's, Toronto, Ontario
  - Toronto General Hospital, Toronto, Ontario
  - Center Hospitalier Universitaire de Montreal, Montreal, Quebec
  - Montreal Heart Institute, Montreal, Quebec
  - Hospital Sacre-Coeur, Montreal, Quebec
  - Institut de Cardiologie Quebec (QC) - Laval, Québec, Quebec
- China (2):
  - Jilin Heart Hospital, Jilin, Changchun
  - Ruijin Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai
- Clinical Hospital Dubrava, Sušak, Zagreb, Croatia
- Al Nas Hospital, Cairo, Qalyubia Governorate, Egypt
- University Hospital Dusseldorf, Düsseldorf, Germany
- G Kuppuswamy Naidu Memorial Hospital (GKNM), Palayam, Tamil Nadu, India
- European Hospital, Via Portuense, Roma, RM, Italy
- Instituto Mexicano del Seguro Social (IMSS), Mexico City, Mexico
- Medical University of Silesia, Katowice, Poland
- Portugal (2):
  - Unidade Local de Saude Lisboa Ocidental (ULSLO), Lisbon
  - Centro Hospitalar e Universitário Sao João, Porto
- Dedinje Cardiovascular Institute, Belgrade, Serbia
- Spain (4):
  - Hospital Clinic de Barcelona (ICCV), Barcelona, L'Eixample
  - Hospital Clínico Universitario Virgen de la Arrixaca, El Palmar, Murcia
  - Hospital del Vinalopó, Alicante
  - Hospital Universitario de Navarra, Pamplona

REFERENCES:
- [Derived] Fremes SE, Marquis-Gravel G, Gaudino MFL, Jolicoeur EM, Bedard S, Masterson Creber R, Ruel M, Vervoort D, Wijeysundera HC, Farkouh ME, Rouleau JL; STICH3C Study Investigators. STICH3C: Rationale and Study Protocol. Circ Cardiovasc Interv. 2023 Aug;16(8):e012527. doi: 10.1161/CIRCINTERVENTIONS.122.012527. Epub 2023 Aug 15. PMID 37582169